CLINICAL TRIAL: NCT05529914
Title: Effects of Myofascial Release and Neuromuscular Training for Pes Anserine Syndrome Associated With Knee Osteoarthritis: A Randomized Control Trial
Brief Title: Effects of Myofascial Release and Neuromuscular Training for Pes Anserine Syndrome Associated With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Rabia Hassan, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHassan
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis; Pes Anserine Bursitis
MeSH Terms: conditions — Osteoarthritis, Knee; Bursitis | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release + Neuromuscular exercises + Cold pack (Experimental)
  Interventions: Other: Myofascial release; Other: Neuromuscular exercises; Other: Cold pack
- Neuromuscular exercises + Cold pack (Active Comparator)
  Interventions: Other: Neuromuscular exercises; Other: Cold pack

INTERVENTIONS:
Other: Myofascial release — It is a type of physical therapy often used to treat myofascial pain syndrome with pressure.
  Arms: Myofascial release + Neuromuscular exercises + Cold pack
Other: Neuromuscular exercises — Exercises commonly utilized in neuromuscular training programs to improve strength, balance , speed and agility. It will comprised of Warm-up, Lunges, Sideways exercises, Wall squats, Weight transfer exercise, Step up & down, Cool-down
Other: Cold pack — Application of cold pack around the patient's body, and covered with dry towel
  Other Names: Cold pack therapy

SUMMARY:
A randomized control trial will be conducted at the outpatient department of Dow Institute of Physical Medicine and Rehabilitation. A sample size of 80 is calculated using PASS version 11 software. The subjects will be first screened and those who fulfill the inclusion criteria, will be asked to fill the consent form. After selection, the participants will be randomly allocated by the help of computer generated randomization sheet, into two groups i.e. experimental and the control group. The group A will be provided with the myofascial release along with the neuromuscular training whereas the group B will only receive the neuromuscular training. Cold pack will be applied to both the groups. The neuromuscular training consists of warm-up phase, lunges, sideways exercises, wall squats, weight transfer exercises, step up and down and the cool down phase. Total 12 sessions of 35 minutes each will be given to all the participants for about 4 weeks on alternate days. Outcome measures will be analyzed by visual analogue scale (VAS) for pain assessment, goniometry for range of motion and the Knee injury and Osteoarthritis Outcome Score (KOOS) to evaluate the functional assessment of the patients at the baseline and the post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and Females both with the age between 40-60 years.
* Patients with unilateral or bilateral knee osteoarthritis with pes anserine syndrome.
* Patients with knee pain more than 3.4 cm on visual analogue scale as minimum cut of value.
* Kellgren and Lawrence grade II and III on radiological findings.
* Duration of knee osteoarthritis more than 3 months (chronic).

Exclusion Criteria:

* Patients with any neurological disorder.
* Knee deformities such as contractures, genu valgum and genu varum.
* Septic knee arthritis.
* History of ligamentous injury or meniscal tear.
* Cancer or any other malignancy or bone tumor.
* Any history of previous lower limb arthroplasty or other knee surgery.
* Comorbid like diabetes mellitus.
* Inflammatory rheumatic disease (R.A).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity on visual analogue scale after four weeks | Baseline and 4 weeks
  The Visual Analogue Scale is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between pains with similar conditions.. It is 0 to 10 cm scale. Patients rate their pain on that scale. Higher the score in centimeter, severe will be the pain experienced.
Change in range of motion assessed with universal goniometer after four weeks | Baseline and 4 weeks
  The Goniometer is an instrument for the precise measurement of range of movement angles in degree , especially one used to measure the angles before and after range of motion.. Increase in the degree of angle suggests increase in range of movement.

SECONDARY OUTCOMES:
Change in functional disability assessed with Knee injury and osteoarthritis outcome score after four weeks. | Baseline and 4 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems regarding functional disability. In consists of total 100 scores. Increase in scores suggests decreased functional disability and decrease in scores suggests increased functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Farhan I Khan, PhD, Study Director — Dow University of Health Sciences
Locations (2):
- Pakistan (2):
  - Dow Institute of Physical Medicine and Rehabilitation, Karachi, Sindh
  - Sindh Institute of Physical Medicine and Rehabilitation, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No